CLINICAL TRIAL: NCT06178315
Title: Randomized Trial of EUS-guided Celiac Plexus Block vs. Sham for Palliation of Pain in Chronic Pancreatitis
Brief Title: EUS-guided Celiac Plexus Block vs. Sham in Chronic Pancreatitis
Acronym: EPOCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orlando Health, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2103069
Record Dates: First submitted 2023-12-08; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic ultrasound-guided celiac plexus block (Active Comparator): EUS-guided celiac plexus block will be performed.
  Interventions: Procedure: EUS-guided celiac plexus block
- Sham (Sham Comparator): Celiac plexus block will not be performed.
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Procedure: EUS-guided celiac plexus block — Under EUS-guidance, celiac plexus block will be performed with injection of bupivacaine and triamcinolone into the area of celiac plexus.
  Arms: Endoscopic ultrasound-guided celiac plexus block
Procedure: Sham procedure — Celiac plexus will not be performed in this arm.
  Arms: Sham

SUMMARY:
The aim of this randomized trial is to assess the efficacy of EUS-CPB in the alleviation of abdominal pain in patients with chronic pancreatitis.

DETAILED DESCRIPTION:
Chronic pancreatitis is a complex fibroinflammatory disease arising from numerous etiological factors and a variety of clinical manifestations. Abdominal pain is the most debilitating complication and can result in significant morbidity and impact on quality of life. Endoscopic ultrasonography (EUS) has been increasingly utilized for celiac plexus block (EUS-CPB), whereby a steroid in combination with a local anesthetic agent are injected into the celiac plexus within the abdominal cavity. The aim of this randomized trial is to assess the efficacy of EUS-CPB in the alleviation of abdominal pain in patients with chronic pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Abdominal pain of at least 3 months duration and a VAS score ≥ 3, with or without the use of narcotic analgesics.
* Diagnosis of chronic pancreatitis on EUS examination, with ≥ 5 features on EUS.
* No other cause of abdominal pain

Exclusion Criteria:

* Age < 18 years.
* History of prior EUS-CPB.
* Use of anticoagulants that cannot be discontinued for the procedure.
* Clinically significant allergy to bupivacaine or triamcinolone.
* Unable to obtain consent for the procedure from either the patient or LAR.
* Intrauterine pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of adequate pain relief | 1 month
  Rate of adequate pain relief in patients with chronic pancreatitis undergoing endoscopic ultrasound-guided celiac plexus block or sham procedure. Adequate pain relief is defined as a 50% reduction in composite pain score from baseline, measured using the Brief Pain Inventory-Short Form, at 1 month post-intervention.

SECONDARY OUTCOMES:
Technical success | Immediately after procedure
  Successful completion of EUS-CPB.
Pain scores measured using Visual Analog Scale. | 3 months
  Pain score measured using the Visual Analog Scale.
Pain scores measured using the Comprehensive Pain Assessment Tool-Short Form. | 3 months
  Pain score measured using the Comprehensive Pain Assessment Tool-Short Form.
Quality of life assessment | 3 months
  Quality of life score measured using the Pancreatitis Quality of Life Instrument.
Opioid analgesic use | 3 months
  Opioid analgesic use measured in morphine equivalent dosage.
Procedure-related adverse events | 3 months
  Any adverse event occurring as a result of endoscopic intervention.
Disease-related adverse events | 3 months
  Any adverse event occurring as a result of underlying chronic pancreatitis.
Hospital admissions for management of chronic pancreatitis. | 3 months
  Number of hospital admissions for management of chronic pancreatitis.
Length of hospitalization in any patient hospitalized | 3 months
  Length of hospitalization in any patient hospitalized with any adverse event or due to chronic pancreatitis.
Rate of cross-over to EUS-CPB in patients initially assigned to the sham group. | 3 months
  Rate of cross-over to EUS-CPB in patients initially assigned to the sham group.
Rate of need for any additional endoscopic, surgical or radiological intervention for chronic pancreatitis. | 3 months
  Rate of need for any additional endoscopic, surgical or radiological intervention for chronic pancreatitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilcox CM, Bang JY, Buxbaum J, Gardner TB, Hawes R, Kedia P, Mardini SH, Muniraj T, Navaneethan U, Oza VM, Tarnasky P, Thakkar S, Waxman I, Varadarajulu S; US Pancreatic Disease Study Group. Effect of endoscopic ultrasound guided celiac plexus block on the palliation of pain in chronic pancreatitis (EPOCH Trial): study protocol for a randomized multicenter sham-controlled trial 1. Trials. 2024 Oct 14;25(1):676. doi: 10.1186/s13063-024-08478-y. PMID 39396987